CLINICAL TRIAL: NCT04215978
Title: Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of the Anti OX40 Agonist Monoclonal Antibody BGB-A445 in Combination With the Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: Safety and Preliminary Effectiveness of BGB-A445 in Combination With Tislelizumab in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-A445-101; 2022-501177-39-00 (EU CTIS Number); CTR20220453 (Other: ChinaDrugTrials)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor; Non Small Cell Lung Cancer; Head and Neck Squamous Cell Carcinoma (HNSCC); Nasopharyngeal Carcinoma (NPC)
Keywords: OX40; PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1a: BGB-A445 Monotherapy (Experimental): Dose Escalation Part A: Participants will receive intravenous (IV) infusion of BGB-A445 in sequential cohorts of approximately 8 increasing dose levels on day 1 of each 21-day cycle
  Interventions: Drug: BGB-A445
- Phase 1a: BGB-A445 + Tislelizumab Combination Therapy (Experimental): Dose Escalation Part B: Participants will receive IV infusion of BGB-A445 in sequential cohorts of approximately 6 increasing dose levels plus 200mg tislelizumab on day 1 of each 21-day cycle
  Interventions: Drug: BGB-A445; Drug: tislelizumab
- Phase 1b:BGB-A445 Monotherapy (Experimental): Dose Expansion Part A: Participants will receive recommended doses of IV BGB-A445 as determined from Phase 1a Dose Escalation; BGB-A445 will be evaluated in two tumor types
  Interventions: Drug: BGB-A445
- Phase 1b: BGB-A445 + Tislelizumab and Chemotherapy Combination Therapy (Experimental): Dose Expansion Part B: Participants will receive recommended dose IV infusion of BGB-A445 plus 200mg tislelizumab and chemotherapy
  Interventions: Drug: BGB-A445; Drug: tislelizumab
- Phase 1b: BGB-A445 Monotherapy (Experimental): Dose Expansion Part C: Participants will receive 1 dose level of BGB-A445
  Interventions: Drug: BGB-A445

INTERVENTIONS:
Drug: BGB-A445 — Administered as specified in the treatment arm
  Other Names: Gimistotug
Drug: tislelizumab — Administered as specified in the treatment arm
  Other Names: BGB-A317
  Arms: Phase 1a: BGB-A445 + Tislelizumab Combination Therapy; Phase 1b: BGB-A445 + Tislelizumab and Chemotherapy Combination Therapy

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BGB-A445 alone and in combination with tislelizumab in participants with advanced solid tumors; and to determine the maximum tolerated dose(s) (MTD) or maximum administered dose(s) (MAD) and recommended Phase 2 doses (RP2D) of BGB-A445 alone and in combination with tislelizumab.

ELIGIBILITY:
Key Inclusion Criteria:

1. Phase 1a (dose escalation): Participants with histologically or cytologically confirmed advanced, metastatic, unresectable solid tumors who have previously received standard systemic therapy or for whom treatment is not available, not tolerated or refused.

1. Enrollment will be limited to participants with advanced solid tumors for which there is clinical evidence of response to T cell based immuno-oncology agents (eg, anti PD 1) or other scientific evidence in support of an immunologically sensitive tumor type.
2. Participant has not received prior therapy targeting OX40 or any other T cell agonist therapy (prior checkpoint inhibitor therapy is allowed)

   2. Phase 1b, the dose expansion phase, aims to include participants in specific tumor type cohorts who do not have access to standard systemic treatment, cannot tolerate it, or it is deemed inappropriate by the investigator. Cohort 1 focuses on non-small cell lung cancer (NSCLC) patients with advanced or metastatic disease, while Cohort 2 involves individuals with recurrent or metastatic head and neck squamous cell cancer (HNSCC). Cohort 3 includes participants with nasopharyngeal carcinoma (NPC), and Cohort 4 is for NSCLC patients with PD-L1 expression of at least 50%. Each cohort has specific eligibility criteria related to prior therapies, tumor characteristics, and treatment-free intervals.

   3. Has at least 1 measurable lesion as defined per RECIST 1.1. The target lesion(s) selected have not been previously treated with local therapy OR the target lesion(s) selected that are within the field of prior local therapy have subsequently progressed as defined by RECIST 1.1 4. Participants should be able to provide tumor tissue sample 5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 and a life expectancy of ≥ 6 months.

   6. Adequate organ function as indicated by the following laboratory values up to first dose of study drug

a. Participants must not have required blood transfusion or growth factor support ≤ 14 days before sample collection for the following:

* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 75 x 10^9/L
* Hemoglobin ≥ 90 g/L

  b. Estimated glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2 determined by the Cockcroft-Gault formula without correction for body surface area (BSA)
* The estimated GFR for participants with renal cell carcinoma must be ≥ 30 mL/min/1.73 m^2 by the Cockcroft-Gault formula

  c. Serum total bilirubin ≤ 1.5 x ULN (< 3 x ULN for participants with Gilbert syndrome) d. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN;
* ≤ 5 x ULN for participants with hepatocellular carcinoma or liver metastases

Key Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled brain metastasis. Participants with equivocal findings or with confirmed brain metastases are eligible for enrollment provided they are asymptomatic and radiologically stable without the need for corticosteroid treatment for at least 4 weeks prior to the first dose of study drug(s)
2. Active autoimmune diseases or history of autoimmune diseases that may relapse or history of life-threatening toxicity related to prior immune therapy, with the following exceptions:

   1. Controlled type 1 diabetes
   2. Hypothyroidism (provided it is managed with hormone-replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, or alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors (requires consultation with the medical monitor prior to enrollment)
3. Any active malignancy ≤ 2 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast)
4. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug(s), with the following exceptions:

   1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption
   3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a nonautoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen)
5. Any major surgical procedure occurring ≤ 28 days before the first dose of study drug(s). If surgical procedure occurs > 28 days, they must have recovered adequately from the toxicity

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants Experiencing Adverse Events (AEs) | Up to 90 days after the last dose of study drug(s) regardless of whether the participant starts a subsequent anticancer therapy
Phase 1a: Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 90 days after the last dose of study drug(s) regardless of whether the participant starts a subsequent anticancer therapy
Phase 1a: Number of Participants Experiencing AEs meeting protocol defined Dose-Limiting Toxicity (DLT) criteria | Up to 90 days after the last dose of study drug(s) regardless of whether the participant starts a subsequent anticancer therapy
Phase 1a: Maximum Tolerated Dose (MTD) of BGB-A445 | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
  The MTD is defined as the highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30%
Phase 1b: RP2D of BGB-A445 when Administered Alone | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1b: Overall Response Rate (ORR) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
  ORR is defined as the proportion of participants who had confirmed complete response Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Phase 1a: Overall Response Rate (ORR) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1a: Duration of Response (DOR) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1a: Disease-Control Rate (DCR) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1a: Serum Concentration of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1a: Serum Concentration of tislelizumab | 60 minutes predose up to 72 hours postdose
Phase 1a: Maximum Observed Plasma Concentration (Cmax) of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1a: Maximum Observed Plasma Concentration (Cmax) of tislelizumab | 60 minutes predose up to 72 hours postdose
Phase 1a: Minimum Observed Plasma Concentration (Cmin) of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1a: Minimum Observed Plasma Concentration (Cmin) of tislelizumab | 60 minutes predose up to 72 hours postdose
Phase 1a: Time to Maximum Plasma Concentration (Tmax) of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1a: Time to Maximum Plasma Concentration (Tmax) of tislelizumab | 60 minutes predose up to 72 hours postdose
Phase 1a: Area Under the Concentration-Time Curve of 0-21 Days (AUC0-21d) of BGB-A445 | 60 minutes predose up to 21 days postdose
Phase 1a: Immunogenic Responses to BGB-A445 as assessed through the detection of antidrug antibodies | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1a: Immunogenic Responses to tislelizumab as assessed through the detection of antidrug antibodies | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1b: Progression-free survival (PFS) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
  Determined from investigator derived tumor assessments as per RECIST 1.1
Phase 1b: Duration of Response (DOR) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1b: Disease-Control Rate (DCR) as Assessed by the Investigator | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first
Phase 1b: Number of Participants Experiencing Adverse Events (AEs) | Up to 90 days after the last dose of study drug(s) regardless of whether the participant starts a subsequent anticancer therapy
Phase 1b: Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 90 days after the last dose of study drug(s) regardless of whether the participant starts a subsequent anticancer therapy
Phase 1b: Serum Concentration of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1b: Maximum Observed Plasma Concentration (Cmax) of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1b: Minimum Observed Plasma Concentration (Cmin) of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1b: Time to Maximum Plasma Concentration (Tmax) of BGB-A445 | 60 minutes predose up to 72 hours postdose
Phase 1b: Area Under the Concentration-Time Curve of 0-21 Days (AUC0-21d) of BGB-A445 | 60 minutes predose up to 21 days postdose
Phase 1b: Immunogenic Responses to BGB-A445 as assessed through the detection of antidrug antibodies | Up to 30 days after the last dose of study drug(s) or before the initiation of a new anticancer treatment, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (30):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - California Cancer Associates for Research & Excellence (cCARE), San Diego, California
  - UPMC Hillman Cancer Center (Univ Of Pittsburgh), Pittsburgh, Pennsylvania
- Australia (7):
  - Blacktown Cancer And Haematology Centre, Blacktown, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (7):
  - Union Hospital Of Tongji Medical College, Huazhong University Of Science And Technology, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Affiliated Zhongshan Hospital Of Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Malaysia (2):
  - University of Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - National Cancer Center (NCC), Goyang-si, Gyeonggi-do
  - Cha Bundang Medical Center, Cha University, Gyeonggido, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
- Taiwan (2):
  - Changhua Christian Hospital, Changhua, NAP
  - National Cheng Kung University Hospital, Tainan
- Thailand (3):
  - King Chulalongkorn Memorial Hospital (Chulalongkorn University), Bangkok
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Srinagarind Hospital (Khon Kaen University), Muang

IPD SHARING:
Plan to Share IPD: Yes